CLINICAL TRIAL: NCT02623491
Title: A Double-Blind, Placebo-Controlled, Randomized, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-55375515 in Healthy Subjects
Brief Title: Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-55375515 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CR108063; 2015-003817-31 (EudraCT Number); 55375515EDI1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-11-18; First posted 2015-12-07 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: JNJ-55375515; Healthy; Placebo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: Single Ascending Dose (SAD) (Experimental): Participants will receive 0.75 milligrams (mg) of JNJ-55375515 (starting dose) or Placebo on Day 1. Dose of the study medication will be escalated sequentially up to a maximum of 200 mg.
  Interventions: Drug: JNJ-55375515; Drug: Placebo
- Part 2: Multiple Ascending Dose (MAD) (Experimental): Participants will receive JNJ-55375515 (at doses determined based on the data from the SAD part) or Placebo from Day 1 to 10.
  Interventions: Drug: JNJ-55375515; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-55375515 — Participants will receive JNJ-55375515 at a starting dose of 0.75 milligrams (mg) and maximum escalated dose will be 200 mg.
Drug: Placebo — Participants will receive matching placebo.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of JNJ-55375515 in healthy participants after administration of single and multiple oral doses.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), double-blind (neither the investigator nor the participants know what treatment the participant is receiving), placebo-controlled (an inactive comparator treatment that has no study drug in it), single center study in healthy male participants and female participants of non-childbearing potential (surgically sterile or post menopausal), aged 18 to 58 years inclusive. This study will consist of two parts; a Single Ascending Dose (SAD) part and a Multiple Ascending Dose (MAD) part. The SAD will consist of 6 escalating dose cohorts. Participants in each cohort will be randomized to receive a single oral administration of JNJ-55375515 or placebo after an overnight fast. The planned doses of JNJ-55375515 range from 0.75 to 100 milligrams (mg). Participants in an additional cohort will be dosed in the fed state to determine the effects of food on the safety, tolerability and pharmacokinetics of JNJ-55375515. An additional optional cohort may be evaluated to further explore the safety, tolerability, pharmacokinetics, and pharmacodynamics of JNJ-55375515, with the maximal dose not exceeding 200 mg. The study duration for participants in the SAD part of the study will be approximately 2 to 5.5 weeks, including eligibility Screening. The MAD will consist of 3 cohorts of 9 participants. Participants will receive once daily oral doses of JNJ-55375515 or placebo for 10 consecutive days. The study duration for participants in the MAD part of this study will be approximately 3 to 7 weeks including the eligibility Screening. The Safety of Participants will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy on the basis of physical and neurological examination, medical history, vital signs, and electrocardiogram (ECG), and have a body mass index of 18-30 kilogram / square meter (kg/m^2) and a body mass of not less than 50 kg.
* Participant must be healthy on the basis of clinical laboratory tests performed at Screening and Day -1.
* Female participants must not be of childbearing potential by either being post-menopausal or permanently sterilized.
* Female participants must not be pregnant.
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol, including contraception.
* Each participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and are willing to participate in the study.

Exclusion Criteria:

* Participant has current, or history of, clinically significant medical or psychiatric illness.
* Participant has any condition for which participation would not be in the best interest of the participant or that could prevent, limit, or confound any protocol specified assessments or the interpretation of the study results.
* Participant has a personal history of, or a first degree relative with a history of, acute angle-closure glaucoma, or participant has significant hyperopia (far-sightedness).
* Participant has a QT corrected according to Fridericia's formula (QTcF) interval greater than (>) 450 msec (male) or >470 msec (female), or has a history of additional risk factors for torsades de pointes.
* Participant has history of vasovagal episodes.
* Participant has history of drug, alcohol, nicotine, or caffeine abuse.
* Participant who is breastfeeding.
* Participant has had major surgery within 12 weeks of Screening, has donated more than 450 milliliters (mL) of blood, or has acute loss of equivalent amount of blood within 90 days of study drug administration.
* Participant has positive fecal occult blood test results at Screening.
* Participant has history of clinically significant drug and/or food allergies.
* Participant has received another investigational drug within 1 month or a period of less than 10 times the drug's half-life, whichever is longer, before the planned first dose of study drug
* Participant is an employee, or family member of an employee, of the study site.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to Day 7 after discharge
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Part 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) | Up to Day 5
  The Tmax is defined as actual sampling time to reach maximum observed concentration.
Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) | Up to Day 5
  The AUC(0-t) is the area under the plasma concentration-time curve from time zero to any time 't'.
Part 1: Elimination Half-Life (t1/2) | Up to Day 5
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Part 1: Maximum Observed Plasma Concentration (Cmax) | Up to Day 5
  The Cmax is the maximum observed concentration.
Part 2: Time to Reach Maximum Observed Plasma Concentration (Tmax) | Up to Day 15
  The Tmax is defined as actual sampling time to reach maximum observed concentration.
Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) | Up to Day 15
  The AUC(0-t) is the area under the plasma concentration-time curve from time zero to any time 't'.
Part 2: Elimination Half-Life (t1/2) | Up to Day 15
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Part 2: Maximum Observed Plasma Concentration (Cmax) | Up to Day 15
  The Cmax is the maximum observed concentration.

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) of JNJ-55375515 | Up to Day 5 in part 1; up to Day 15 in part 2
  The maximum tolerated dose is defined as the dose below the dose at which 2 or more subjects receiving the same dose of active study drug experience the same dose-limiting toxicity or have the same severe adverse event, or below the level at which the Investigator and Sponsor agree that an unacceptable dose-limiting toxicity has occurred in a single subject treated with active study drug.
Part 1: The Effect of Food on the Number of Adverse Events | Baseline up to Day 5
Part 1: The Effect of Food on Maximum Observed Plasma Concentration (Tmax) | Baseline up to Day 5
Part 1: The Effect of Food on Maximum Observed Plasma Concentration (Cmax) | Baseline up to Day 5
Part 1: The Effect of Food on Elimination Half-Life (t1/2) | Baseline up to Day 5
Part 1: The Effect of Food on Area Under the Plasma Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) | Baseline up to Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium